CLINICAL TRIAL: NCT04397133
Title: The Optimal Treatment Duration for Inspiratory Muscle Strengthening Exercises in Stroke Patients: A Double-blind Randomised Controlled Trial
Brief Title: The Optimal Treatment Duration for Inspiratory Muscle Strengthening Exercises in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Collaborators: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IstPMRTRH-IMT-H
Record Dates: First submitted 2019-11-11; First posted 2020-05-21 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Stroke, Complication; Respiratory Complication
Keywords: Breathing exercises; Cerebrovascular disease; Muscle strength; Rehabilitation; Stroke
MeSH Terms: conditions — Stroke; Cerebrovascular Disorders

STUDY DESIGN:
Intervention Model Description: three armed study with two interventions and one control group intervention group 1: inspiratory muscle training applied for 4 week intervention group 2: inspiratory muscle training applied for 8 week control group : will get sham intervention
Who Masked: Investigator, Outcomes Assessor
Masking Description: the assessor who will investigate the results and the investigator who will perform the MIP and 6-minutes walking test will be blinded to the randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- intervention 1 (Experimental): in this group patients will get 4 week of inspiratory muscle training exercise 30 minutes every weekday ( 15 minutes of two session in each day)
  Interventions: Other: inspiratory muscle training
- intervention 2 (Experimental): in this group patients will get 8 week of inspiratory muscle training exercise 30 minutes every weekday ( 15 minutes of two session in each day)
  Interventions: Other: inspiratory muscle training
- control group (Sham Comparator): this group will get sham intervention with 0 to 5 cmH2O resistance
  Interventions: Other: sham intervention

INTERVENTIONS:
Other: inspiratory muscle training — inspiratory muscle training will be done with Philips Respironics Threshold IMT device starting with resistance of % 50 of MIP value
  Arms: intervention 1; intervention 2
Other: sham intervention — in these group the patients will get sham intervention with Philips Respironics Threshold IMT device
  Arms: control group

SUMMARY:
The first aim of this study is if there is any difference between 4 or 8 weeks of inspiratory muscle training ( IMT ) exercises groups and control groups in stroke survivors. The secondary aims of this study is if there is any difference in walking capacity (in 8th, 12th, 24th weeks) and pulmonary complications (pneumonia incidences) in long term follow-ups (6 months) in these aforementioned groups

DETAILED DESCRIPTION:
Stroke is one of the leading causes of death and disability. It is not only because of loss of extremity motions but also loss of inspiratory muscle strength. In this study we aimed to determine the optimum duration for inspiratory muscle training exercises for stroke survivors since there is not enough data about it in the literature.

The study will include at least 54 patients in total and 18 in each groups ( two intervention and one control) . The patients will be evaluated for angina, chronic obstructive pulmonary disease, congestive heart disease; in these conditions the patients will be excluded from the study. Also in first examinations we will evaluate the maximal inspiratory pressure (MIP) of patients, of them the ones with MIP measurements above 80 mmH2O will also be excluded since it is the expected value in normal people.

After admission and randomizing the patients, baseline measurements of MIP, 6-minutes walking test will be done. In intervention groups the patients will get 30 minutes of inspiratory muscle training exercises ( 15 minutes of two session each day) with threshold IMT device every weekday. And in control group, the patients will get sham intervention for 8 weeks. The MIP and 6-minutes walking test will be done in 8th,12th and 24th weeks. And also in 24th week we will record the pneumonia incidence if occured.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic/ hemorrhagic stroke
* Stroke duration> 3 months
* Age> 18 years old
* Baseline maximal inspiratory pressure below 80 cmH2O

Exclusion Criteria:

* Cognitive deficiency
* Facial paralysis
* Chronic obstructive pulmonary disease
* Congestive heart disease
* Myocardial infarction in last three months
* Angina pectoris

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-12-23 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
The change in maximal inspiratory pressure | Baseline and week 8,12, 24
  Measured with MicroRPM (respiratory pressure meter) pressurometer device orally

SECONDARY OUTCOMES:
The change in walking capacity | Baseline and week 8,12, 24
  The change in walking capacity wil be measured with Six Minute Walk Test
Pneumonia incidence | Week 24
  Number of participants with Pneumonia will be determined at week 24

CONTACTS AND LOCATIONS:
Overall Officials: Yunus Emre Doğan, MD, Principal Investigator — Istanbul Physical Medicine Rehabilitation Traning and Research Hospital; Burak Kütük, MD, Principal Investigator — Istanbul Physical Medicine Rehabilitation Traning and Research Hospital
Locations (1):
- Istanbul Physical Medicine Rehabilitation Traning and Research Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Pollock RD, Rafferty GF, Moxham J, Kalra L. Respiratory muscle strength and training in stroke and neurology: a systematic review. Int J Stroke. 2013 Feb;8(2):124-30. doi: 10.1111/j.1747-4949.2012.00811.x. Epub 2012 May 9. PMID 22568454
- [Background] Britto RR, Rezende NR, Marinho KC, Torres JL, Parreira VF, Teixeira-Salmela LF. Inspiratory muscular training in chronic stroke survivors: a randomized controlled trial. Arch Phys Med Rehabil. 2011 Feb;92(2):184-90. doi: 10.1016/j.apmr.2010.09.029. PMID 21272713
- [Background] Guillen-Sola A, Messagi Sartor M, Bofill Soler N, Duarte E, Barrera MC, Marco E. Respiratory muscle strength training and neuromuscular electrical stimulation in subacute dysphagic stroke patients: a randomized controlled trial. Clin Rehabil. 2017 Jun;31(6):761-771. doi: 10.1177/0269215516652446. Epub 2016 Jun 7. PMID 27271373
- [Background] Billinger SA, Coughenour E, Mackay-Lyons MJ, Ivey FM. Reduced cardiorespiratory fitness after stroke: biological consequences and exercise-induced adaptations. Stroke Res Treat. 2012;2012:959120. doi: 10.1155/2012/959120. Epub 2011 Aug 14. PMID 21876848
- [Background] Sutbeyaz ST, Koseoglu F, Inan L, Coskun O. Respiratory muscle training improves cardiopulmonary function and exercise tolerance in subjects with subacute stroke: a randomized controlled trial. Clin Rehabil. 2010 Mar;24(3):240-50. doi: 10.1177/0269215509358932. Epub 2010 Feb 15. PMID 20156979
- [Background] Katzan IL, Cebul RD, Husak SH, Dawson NV, Baker DW. The effect of pneumonia on mortality among patients hospitalized for acute stroke. Neurology. 2003 Feb 25;60(4):620-5. doi: 10.1212/01.wnl.0000046586.38284.60. PMID 12601102